CLINICAL TRIAL: NCT02095873
Title: Dietary Inducers of Glyoxalase-1 for Prevention and Early-stage Alleviation of Age Related Health Disorders Through Functional Foods.
Brief Title: Healthy Aging Through Functional Food
Acronym: HATFF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Warwick (Other)
Collaborators: Technology Strategy Board, United Kingdom (Other); Unilever R&D (Industry)
Responsible Party: Principal Investigator, Professor Paul J. Thornalley, Professor, University of Warwick
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PJT_HATFF; TSB101129 (Other: University of Warwick)
Record Dates: First submitted 2014-03-18; First posted 2014-03-26 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Glucose Intolerance; Aortic Stiffness; Vasodilation
Keywords: Oral glucose tolerance test; Flow mediated dilatation; Aortal pulse wave velocity; Finger-fold capillary density by capillaroscopy
MeSH Terms: conditions — Glucose Intolerance; Aneurysm | interventions — Lactoylglutathione Lyase; Resveratrol; hesperetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glo1-inducer then placebo (Experimental): Glyoxalase 1 Inducer (8 weeks), then washout (6 weeks), then Placebo (8 weeks).
  Interventions: Dietary Supplement: Glyoxalase 1 (Glo1) inducer; Dietary Supplement: Placebo
- Placebo then Glo1-inducer (Experimental): Placebo (8 weeks), then washout (6 weeks), then Glyoxalase 1 Inducer (8 weeks).
  Interventions: Dietary Supplement: Glyoxalase 1 (Glo1) inducer; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glyoxalase 1 (Glo1) inducer — Dietary bioactive
  Other Names: trans-resveratrol, 90 mg + hesperetin, 120 mg (combination)
Dietary Supplement: Placebo — Mannitol, 108 mg

SUMMARY:
The purpose of this study is to determine whether dietary inducers of glyoxalase 1 are effective in improving metabolic and vascular health.

DETAILED DESCRIPTION:
The aim of the study is to evaluate dietary inducers of glyoxalase 1 for effects on metabolic and vascular health in overweight volunteers at risk of developing type 2 diabetes. The research objectives are:

(i) To evaluate dietary inducers of glyoxalase 1 for effects on markers of glucose metabolism during an oral glucose tolerance test (oGTT), (ii) To evaluate dietary inducers of glyoxalase 1 for effects on vascular function on three levels, using finger fold capillary density by capillaroscopy (FFCD), arterial stiffness by aortal pulse wave velocity (aPWV) and flow mediated dilatation (FMD); and effects on metabolic and pro-inflammatory markers in circulating blood and urine.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 - 40 kg/m2 (>23 kg/m2 for Asians), with normal, impaired fasting or impaired postprandial glucose.
* No other relevant morbidities.
* Women will be preferably post-menopausal.

Exclusion Criteria:

* Severe hypertriglyceridemia.
* Uncontrolled hypertension, cardiovascular disease, relevant renal or hepatic disease, diabetes, and other relevant morbidity.
* Excess alcohol consumption, smoking, acute pharmacological treatment with drugs affecting glucose metabolism such as steroids and antibiotics.
* Anticoagulants.
* Intake of herbal remedies.
* Food allergies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Thornalley, BSc PhD, Study Chair — University of Warwick; Martin O Weickert, MD, Principal Investigator — University Hospitals Coventry & Warwickshire NHS Trust
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust (UHCW), Coventry, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Xue M, Rabbani N, Momiji H, Imbasi P, Anwar MM, Kitteringham N, Park BK, Souma T, Moriguchi T, Yamamoto M, Thornalley PJ. Transcriptional control of glyoxalase 1 by Nrf2 provides a stress-responsive defence against dicarbonyl glycation. Biochem J. 2012 Apr 1;443(1):213-22. doi: 10.1042/BJ20111648. PMID 22188542
- [Background] Rabbani N, Thornalley PJ. Dicarbonyl stress in cell and tissue dysfunction contributing to ageing and disease. Biochem Biophys Res Commun. 2015 Mar 6;458(2):221-6. doi: 10.1016/j.bbrc.2015.01.140. Epub 2015 Feb 7. PMID 25666945
- [Result] Xue M, Weickert MO, Qureshi S, Kandala NB, Anwar A, Waldron M, Shafie A, Messenger D, Fowler M, Jenkins G, Rabbani N, Thornalley PJ. Improved Glycemic Control and Vascular Function in Overweight and Obese Subjects by Glyoxalase 1 Inducer Formulation. Diabetes. 2016 Aug;65(8):2282-94. doi: 10.2337/db16-0153. Epub 2016 May 11. PMID 27207552

RESULTS

PARTICIPANT FLOW:
Groups:
- Glyoxalase 1 Inducer First, Then Placebo: Glyoxalase 1 inducer (capsule, 90 mg trans-resveratrol & 120 mg hesperetin combination) once daily, 8 weeks; then Placebo (excipient: Mannitol, 108 mg) once daily, 8 weeks.
- Placebo Then Glyoxalase 1 Inducer: Placebo (excipient: Mannitol, 108 mg), once daily, 8 weeks; then Glyoxalase 1 inducer (capsule, 90 mg trans-resveratrol & 120 mg hesperetin combination) once daily, 8 weeks.
Period: First Intervention (8 Weeks)
Arm/Group | Glyoxalase 1 Inducer First, Then Placebo | Placebo Then Glyoxalase 1 Inducer
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Glyoxalase 1 Inducer First, Then Placebo | Placebo Then Glyoxalase 1 Inducer
Started | 15 | 16
Completed | 13 | 16
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Glyoxalase 1 Inducer Then Placebo: Glyoxalase 1 inducer (90 mg trans-resveratrol & 120 mg hesperetin), once daily, 8 weeks; then Placebo (excipient: 108 mg mannitol), once daily, 8 weeks.
- Placebo Then Glyoxalase 1 Inducer: Placebo (excipient: 108 mg mannitol), once daily, 8 weeks; then Glyoxalase 1 inducer (90 mg trans-resveratrol & 120 mg hesperetin), once daily, 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Glyoxalase 1 Inducer Then Placebo | Placebo Then Glyoxalase 1 Inducer | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12) | 44 (13) | 45 (13)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Oral Glucose Tolerance Test (oGGT)
Description: A standard 75 g glucose oGTT will be performed, as routinely used in clinical practice. Participants will be instructed to eat carbohydrate rich diet (> 150 g/day) for at least three days before the test, followed by an overnight fast. Participants will be instructed to have comparable macronutrient composition of the dinner before the respective study days in the metabolic unit. During the oGTT both capillary and venous blood samples will be collected after 0, 15, 30, 60, 90 and 120 min. To minimize the inconvenience of repeated blood tests during the oGTT, a venous cannula will be inserted, under sterile conditions, prior to the test, for blood sampling.
Time Frame: Week 0 and Week 8 (first intervention); Week 14 and Week 22 (second intervention)
Population: Highly overweight/obese (BMI>27.5 kg/m2) subgroup, based on subject BMI at study entry.
Measure: Mean (Standard Error); unit: mM h
Groups:
- Glyoxalase 1 Inducer: Glyoxalase 1 inducer (90 mg trans-resveratrol & 120 mg hesperetin), once daily, 8 weeks.
- Placebo: Placebo (excipient: 108 mg mannitol), capsule, once daily, 8 weeks.
Arm/Group | Glyoxalase 1 Inducer | Placebo
Number analyzed (Participants) | 20 | 20
mM h
  Baseline | 10.8 (0.7) | 11.0 (0.7)
  Post-8 weeks treatment | 9.9 (0.6) | 10.6 (0.6)

2. Secondary Outcome: Finger-fold Capillary Density by Capillaroscopy
Description: After 20 min seated at rest, measurements are made with the subject seated and the left hand at heart level. Nail-fold capillaries in the dorsal skin of the third finger are visualized using a stereo microscope linked to a monochrome digital camera. Capillary density is defined as the number of capillaries per mm2 of nail-fold skin and is computed as the mean of 4 measurements.
Time Frame: Week 0 and Week 8 (first intervention); Week 14 and Week 22 (second intervention)
Population: All subjects with where baseline and post-8 treatment data were obtained.
Measure: Median (Inter-Quartile Range); unit: number of capillaries per mm2
Groups:
- Glyoxalase 1 Inducer: Glyoxalase 1 inducer (capsule, 90 mg trans-resveratrol & 120 mg hesperetin combination) once daily, 8 weeks.
- Placebo: Placebo (excipient: Mannitol, 108 mg), once daily, 8 weeks.
Arm/Group | Glyoxalase 1 Inducer | Placebo
Number analyzed (Participants) | 28 | 24
number of capillaries per mm2
  Baseline | 115 [90 to 140] | 119 [107 to 164]
  Post-8 weeks treatment | 125 [88 to 169] | 128 [104 to 149]

3. Secondary Outcome: Flow-mediated Dilatation (FMD)
Description: Brachial artery FMD will be assessed. Ultrasound imaging of the brachial artery will be performed. Percent FMD will be calculated using the averaged minimum mean brachial artery diameter at baseline compared to the largest mean values obtained after either release of the forearm occlusion.
Time Frame: Week 0 and Week 8 (first intervention); Week 14 and Week 22 (second intervention)
Population: All subjects completing the study per protocol
Measure: Median (Inter-Quartile Range); unit: percentage of baseline value
Arm/Group | Glyoxalase 1 Inducer | Placebo
Number analyzed (Participants) | 29 | 29
percentage of baseline value
  Baseline | 0.17 [0.10 to 0.35] | 0.18 [0.07 to 0.49]
  Post-8 weeks treatment | 0.12 [0.06 to 0.31] | 0.26 [0.07 to 0.47]

4. Other Pre Specified Outcome: Aortal Pulse Wave Velocity (aPWV)
Description: Aortal pulse wave velocity is measured by a non-invasive oscillometric device.
Time Frame: Week 0 and Week 8 (first intervention); Week 14 and Week 22 (second intervention)
Population: Subjects for which PWV data were obtained at baseline and post 8-weeks treatment.
Measure: Median (Inter-Quartile Range); unit: m/s
Arm/Group | Glyoxalase 1 Inducer | Placebo
Number analyzed (Participants) | 13 | 12
m/s
  Baseline | 7.9 [7.1 to 8.8] | 8.3 [7.4 to 9.2]
  Post-8 weeks treatment | 8.0 [7.1 to 10.0] | 8.5 [7.5 to 9.0]

ADVERSE EVENTS:
Time Frame: From baseline to study completion: 8 weeks Glo1-inducer, 6 weeks washout then 8 weeks placebo; or 8 weeks placebo, 6 weeks washout then 8 weeks Glo1-inducer.
Description: All potential clinical adverse effects were monitoring including nausea, loss of appetite, gastrointestinal side effects and other symptoms. Clinical chemistry and haematological assessments were also made.
Groups:
- Glo1-inducer Then Placebo: Glyoxalase 1 inducer: capsule, 90 mg trans-resveratrol & 120 mg hesperetin, once daily for 8 weeks; then 6-weeks washout; then placebo capsule (mannitol, 210 mg), once daily for 8 weeks.
- Placebo Then Glo1-inducer: Placebo capsule (mannitol, 210 mg), once daily for 8 weeks; then 6-weeks washout; then Glyoxalase 1 inducer: capsule, 90 mg trans-resveratrol & 120 mg hesperetin, once daily for 8 weeks.
Arm/Group | Glo1-inducer Then Placebo | Placebo Then Glo1-inducer
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes